CLINICAL TRIAL: NCT03907969
Title: A Phase I/IIa, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Ascending Doses of AZD7648 Monotherapy or in Combination With Either Cytotoxic Chemotherapies or Novel Anti-Cancer Agents in Patients With Advanced Malignancies
Brief Title: A Clinical Trial to Evaluate AZD7648 Alone and in Combination With Other Anti-cancer Agents in Patients With Advanced Cancers.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9170C00001; 2018-003688-73 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-04-09 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Advanced Malignancies
Keywords: Safety,; Pharmacokinetics,; Pegylated liposomal doxorubicin,; Dose finding
MeSH Terms: interventions — AZD7648; 1-dodecylpyridoxal; liposomal doxorubicin

STUDY DESIGN:
Masking Description: This is an open-label study; there will be no blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Core Module: AZD7648 Monotherapy (Experimental): AZD7648 will be administered orally on an empty stomach
  Interventions: Drug: AZD7648
- Combination Module 1: AZD7648 + PLD (Experimental): AZD7648 will be administered in combination with Pegylated liposomal doxorubicin (PLD)
  Interventions: Drug: AZD7648; Drug: PLD

INTERVENTIONS:
Drug: AZD7648 — Core: AZD7648 will be administered orally
Drug: PLD — The starting dose of PLD is 40 mg/m^2, administered by intravenous infusion once every 4 weeks, for a maximum of 6 cycles
  Other Names: DOXIL, Caelyx
  Arms: Combination Module 1: AZD7648 + PLD

SUMMARY:
This is a modular Phase I/IIa, open-label, multi-centre, study of AZD7648 administered orally, either as a monotherapy, or in combination with either cytotoxic chemotherapies or novel anti-cancer agents in participants with advanced malignancies.

DETAILED DESCRIPTION:
The modular design allows for an escalation of the dose of AZD7648 alone or in combination with either cytotoxic chemotherapies or novel anti-cancer agents, with intensive safety monitoring to ensure the safety of the participants.

The study consists of 2 modules each evaluating the safety and tolerability of AZD7648 monotherapy or with a specific combination partner.

Core module of the study is dose escalation (Part A) of AZD7648 monotherapy, administered orally, in participants with advanced solid tumours.

Combination module 1 has 2 study parts: Part A consisting of dose escalation cohorts and Part B, a safety and proof of concept Phase IIa expansion. A Safety Review Committee will review evaluable participants at each cohort and assess if the study should progress to Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to give signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
2. Participant must be at least 18 years of age, at the time of signing the ICF.
3. Participants must have histological or cytological confirmation of advanced malignancy considered to be suitable for study treatment.
4. Eastern cooperative oncology group performance status 0-1.
5. Life expectancy greater than 12 weeks.
6. Progressive cancer at the time of study entry.
7. Pharmacodynamics expansion cohorts: Participants must have at least 1 tumour suitable for biopsy and consent to having biopsies collected.
8. Negative pregnancy test (urine or serum) prior to start of dosing for women of childbearing potential.
9. Female participants must be post-menopausal, surgically sterile, or using an acceptable method of contraception for the duration of the study (from the time they sign consent) and for 12 weeks after the last dose of study treatment to prevent pregnancy.
10. For the duration of the study (from the time they sign consent) and for 12 weeks after the last dose of study treatment, sexually active male participants must be willing to use contraception.

Post-menopausal is defined as:

* No menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy). However in the absence of 12 months of amenorrhea, a FSH measurement is insufficient.
* Radiation-induced oophorectomy with last menses greater than 12 months ago.
* Chemotherapy-induced menopause with greater than 12 month interval since last menses.
* Surgical sterilisation.

Exclusion Criteria:

1. Any unresolved toxicities from prior therapy common terminology criteria for adverse event (CTCAE) Grade ≥2 (with the exception of alopecia).
2. Spinal cord compression or brain metastases unless definitively treated, asymptomatic, stable and not requiring steroids for at least 4 weeks.
3. As judged by the Investigator, any evidence of severe or uncontrolled medical conditions including but not limited to:

   • Uncontrolled diabetes mellitus, uncontrolled seizures, active infection requiring systemic antibiotics, antifungal or antiviral drugs, severe chronic obstructive pulmonary disease, severe Parkinson's disease, active inflammatory bowel disease, psychiatric condition, active bleeding diatheses, renal transplant, or active infection including any participant with active hepatitis B, hepatitis C or human immunodeficiency virus.
4. Any other malignancy which has been active or treated within the past 3 years, with the exception of in situ cancer of the cervix, non-melanoma skin cancer, ductal carcinoma in situ, Stage 1 Grade 1 endometrial carcinoma, or other solid tumours including lymphomas curatively treated with no evidence of disease for ≥5 years.
5. Refractory nausea and vomiting or unable to swallow and retain oral medication, chronic gastrointestinal diseases or previous bowel resection with clinically significant sequelae that would preclude adequate absorption of AZD7648, gastrointestinal symptoms CTCAE Grade >1, history of gastrointestinal ulceration and gastrointestinal haemorrhage within 6 months of first study drug administration.

6 Receiving or having received anti-cancer treatment within the following periods prior to the first dose of investigational product:

(a) Cytotoxic treatment: 3 weeks, (b) Non-cytotoxic drugs: including small molecule investigational products: 3 weeks or 5 half-lives (whichever is longest), (c) Biological products including investigational immuno-oncology agents: 4 weeks, (d) Radiation with a limited field for palliation: 1 week (3 months for radiation to the abdomen or pelvis), (e) Radiation to >30% of the bone marrow or with a wide field: 4 weeks, (f) Lung radiation: 60 days, (g) Major surgery: 4 weeks; minor surgery or biopsy: 1 week 7. During the 4 weeks prior to the first dose, receiving corticosteroids at a dose of >10 mg prednisone/day or equivalent for any reason. Ongoing low dose steroids for longer than 3 months (excluding inhalational, nasal, creams, lotions, and gels) are not allowed.

8. Receiving or having received concomitant medications, herbal supplements and/or foods known to significantly modulate CYP3A4 activity.

9. Prior exposure to a deoxyribonucleic acid-pharmacokinetics inhibitor or hypersensitivity to any excipient of the product.

10. Cardiac dysfunction as defined by any of the following within 6 months of study entry:

(a) Acute myocardial infarction, (b) New York Heart Association Class II/III/IV heart failure, (c) Unstable angina, (d) Unstable cardiac arrhythmias 11. Any of the following cardiac criteria:

(a) Known reduced left ventricular ejection fraction below the institutional lower limit of normal, (b) Mean resting corrected QT interval (QTc) >470 milliseconds obtained from 3 electrocardiograms in 24 hours using the Fridericia formula, (c) Any factors that increase the risk of QTc prolongation or arrhythmic events such as hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age 12. Inadequate hematological or organ function 13. Involvement in the planning and/or conduct of the study. 14. Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.

15. Previous enrolment in the present study. 16. For female participant only: currently pregnant or breast-feeding. 17. For food effect cohort only: insulin dependent diabetes. 18. History and/or presence of coronavirus disease 2019.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Timothy Yap, Principal Investigator — MD Anderson Cancer Center, 1400 Holcombe Blvd. Houston, Texas, 77030
Locations (4):
- United States (2):
  - Research Site, New Haven, Connecticut
  - Research Site, Houston, Texas
- United Kingdom (2):
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Goldberg FW, Finlay MRV, Ting AKT, Beattie D, Lamont GM, Fallan C, Wrigley GL, Schimpl M, Howard MR, Williamson B, Vazquez-Chantada M, Barratt DG, Davies BR, Cadogan EB, Ramos-Montoya A, Dean E. The Discovery of 7-Methyl-2-[(7-methyl[1,2,4]triazolo[1,5-a]pyridin-6-yl)amino]-9-(tetrahydro-2H-pyran-4-yl)-7,9-dihydro-8H-purin-8-one (AZD7648), a Potent and Selective DNA-Dependent Protein Kinase (DNA-PK) Inhibitor. J Med Chem. 2020 Apr 9;63(7):3461-3471. doi: 10.1021/acs.jmedchem.9b01684. Epub 2020 Jan 15. PMID 31851518
- See also: Protocol redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9170C00001&attachmentIdentifier=7da79a41-146a-47d9-ad55-18435eb11ac4&fileName=D9170C00001_PXL_241785_CSP_English_Redacted_final_3.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9170C00001&attachmentIdentifier=f984e580-b359-43a6-b89f-8cf5124f3ac5&fileName=D9170C00001_PXL_241785_SAP_redacted_Redacted_Final_3.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9170C00001&attachmentIdentifier=03124a4e-c667-4686-b36b-860768565776&fileName=D9170C00001-PXL241785-CSR-Synopsis-redacted_Redacted_Final.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 patients were enrolled at two sites in the United States and three sites in the United Kingdom from 09 October 2019 to 07 December 2022.
Pre-assignment Details: Patients who met the inclusion and none of the exclusion criteria were enrolled to the study. This study consisted of a screening period of 28 days. All the study assessments were performed as per schedule of assessment.
Groups:
- Cohort 1: AZD7648 Dose A (Monotherapy): Patients received single dose A of AZD7648, and after a washout period patients received multiple continuous dosing of dose A of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 2: AZD7648 Dose A1 (Monotherapy): Patients received single dose A1 of AZD7648, and after a washout period patients received multiple continuous dosing of dose A of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 3: AZD7648 Dose B1 (Monotherapy): Patients received single dose B1 of AZD7648, and after a washout period patients received multiple continuous dosing of dose B1 of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 4: AZD7648 Dose C1 (Monotherapy): Patients received single dose C1 of AZD7648, and after a washout period patients received multiple continuous dosing of dose C1 of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 5: AZD7648 Dose D1 (Monotherapy): Patients received single dose D1 of AZD7648, and after a washout period patients received multiple continuous dosing of dose D1 of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 6: AZD7648 Dose E1 (Monotherapy): Patients received single dose E1 of AZD7648, and after a washout period patients received multiple continuous dosing of dose E1 of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 7: AZD7648 Dose F1 (Monotherapy): Patients received single dose F1 of AZD7648, and after a washout period patients received multiple continuous dosing of dose F1 of AZD7648 in 28-day cycle regimen orally on an empty stomach.
- Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy): Patients received continuous dosing of dose C1 of AZD7648 orally on an empty stomach. In combination of AZD7648 patients also received PLD of 40 mg/m^2, administered by intravenous (IV) infusion once every 4 weeks.
- Cohort 1: AZD7648 Dose C + PLD (Combination Therapy): Patients received single dosing of dose C of AZD7648 orally on an empty stomach. In combination of AZD7648 patients also received PLD of 40 mg/m^2, administered by IV infusion once every 4 weeks.
- Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy): Patients received single dosing of dose C2 of AZD7648 orally on an empty stomach. In combination of AZD7648 patients also received PLD of 40 mg/m^2, administered by IV infusion once every 4 weeks.
- Cohort 3: AZD7648 Dose X + PLD (Combination Therapy): Patients received single dosing of dose X of AZD7648 orally on an empty stomach. In combination of AZD7648 patients also received PLD of 40 mg/m^2, administered by IV infusion once every 4 weeks.
Period: Monotherapy Part A
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Started | 1 | 1 | 1 | 1 | 3 | 4 | 3 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Combination Therapy Part A
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other than specified main reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least 1 dose of any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 3 | 2 | 2 | 5 | 7 | 30
Age, Customized [Mean (Standard Deviation); unit: Years] | NA (NA) — Not calculable due less number of participants | NA (NA) — Not calculable due less number of participants | NA (NA) — Not calculable due less number of participants | NA (NA) — Not calculable due less number of participants | 64.3 (6.35) | 60.3 (8.18) | 51.3 (2.08) | NA (NA) — Not calculable due less number of participants | NA (NA) — Not calculable due less number of participants | 56.6 (10.16) | 61.7 (16.18) | 60.20 (10.20)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  All | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 11
  Male | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 4
  Female | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 3 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Other | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 0 | 0 | 0 | 2 | 14
  Race: White | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 5 | 5 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Area Under Plasma Concentration-time Curve From Zero to Infinity (AUCinf)
Description: The AUCinf of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents.
Time Frame: Monotherapy and Combination therapy: Cycle 0 Day 1 Pre-dose to 72 hours post-dose [each cycle is 28 days]
Population: All patients who received at least 1 dose of any study treatment and had at least 1 reportable post first dose concentration without any protocol deviations that might have affected pharmacokinetic (PK).
Measure: Geometric Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 4 | 7
h*nmol/L | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 25180 (48.76) | 29680 (19.72) | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 3826 (55.72) | 5539 (52.04)

2. Secondary Outcome: Area Under the Plasma Concentration-curve From Zero to the Last Quantifiable Concentration (AUClast)
Description: The AUClast of AZD7648, following a single dose, when given orally as monotherapy and in combination with anti-cancer agents.
Time Frame: Monotherapy and Combination therapy: Cycle 0 Day 1 Pre-dose to 72 hours post-dose (each cycle is 28 days)
Population: All patients who received at least 1 dose of any study treatment and had at least 1 reportable post first dose concentration without any protocol deviations that might have affected PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 3 | 2 | 2 | 4 | 7
h*nmol/L | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 24940 (49.04) | 29540 (19.64) | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 3798 (55.78) | 5509 (52.19)

3. Secondary Outcome: Area Under Plasma Concentration-time Curve in the Dosing Interval τ (AUCτ)
Description: The AUCτ of AZD7648, at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents.
Time Frame: Monotherapy and Combination therapy: Cycle 0 Day 1 Pre-dose to 72 hours post-dose (each cycle is 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Groups:
- AZD7648 + PLD Dose X (Combination Therapy): Patients received single dosing of dose B of AZD7648 orally on an empty stomach. In combination of AZD7648 patients also received PLD of 40 mg/m^2, administered by IV infusion once every 4 weeks.
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | AZD7648 + PLD Dose X (Combination Therapy)
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1
h*nmol/L | NA (NA) — Mean cannot be calculated due to low number participant. |  | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. |  |  |  | NA (NA) — Mean cannot be calculated due to low number participants. | NA (NA) — Mean cannot be calculated due to low number participants. | NA (NA) — Mean cannot be calculated due to low number participants.

4. Secondary Outcome: Maximum Observed Plasma (Peak) Drug Concentration After Single Dose and Multiple Doses (Cmax)
Description: The Cmax of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents.
Time Frame: Monotherapy: Cycle 0 Day 1 Pre-dose to 72 hours post-dose, Cycle 1 Day 8 Pre-dose to 12 hours post dose; Combination therapy: Cycle 0 Day 1 Pre-dose to 12 hours post dose and Cycle 1 Days 7, 8 Pre-dose to 8 hours post dose (each cycle is 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 3 | 2 | 2 | 4 | 7
nmol/L
  Cycle 0 Day 1 | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 2463 (56.72) | 4026 (13.97) | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 376.8 (27.66) | 754.2 (34.29)
  Cycle 1 Day 7 Cycle 1 Day 8: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 0 | 1 | 5
  Cycle 1 Day 7 Cycle 1 Day 8 | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 5426 (12.75) | NA (NA) — Mean cannot be calculated due to low number participant. |  | NA (NA) — Mean cannot be calculated due to low number participant. | 944.9 (62.85)

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: The tmax of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 3 | 3 | 2 | 2 | 5 | 7
Hours
  Cycle 0 Day 1 | NA [1.08 to 1.08] — Median cannot be calculated due to low number participants. | NA [2.17 to 2.17] — Median cannot be calculated due to low number participants. | NA [1.00 to 1.00] — Median cannot be calculated due to low number participants. | NA [1.03 to 1.03] — Median cannot be calculated due to low number participants. | NA [2.07 to 9.00] — Median cannot be calculated due to low number participants. | 2.050 [2.03 to 2.13] | 2.033 [1.08 to 2.07] | NA [1.07 to 2.08] — Median cannot be calculated due to low number participants. | NA [1.08 to 2.08] — Median cannot be calculated due to low number participants. | 3.058 [1.95 to 8.07] | 1.150 [0.68 to 2.17]
  Cycle 1 Day 7 Cycle 1 Day 8: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 2 | 3 | 2 | 0 | 1 | 5
  Cycle 1 Day 7 Cycle 1 Day 8 | NA [1.12 to 1.12] — Median cannot be calculated due to low number participants. | NA [2.07 to 2.07] — Median cannot be calculated due to low number participants. | NA [1.05 to 1.05] — Median cannot be calculated due to low number participants. | NA [2.00 to 2.00] — Median cannot be calculated due to low number participants. | NA [2.00 to 2.00] — Median cannot be calculated due to low number participants. | NA [2.07 to 2.15] — Median cannot be calculated due to low number participants. | 2.167 [2.10 to 2.42] | NA [1.08 to 2.00] — Median cannot be calculated due to low number participants. |  | NA [2.03 to 2.03] — Median cannot be calculated due to low number participants. | 1.100 [1.00 to 2.20]

6. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz)
Description: The t½λ of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents.
Time Frame: Monotherapy and Combination therapy: Cycle 0 Day 1 Pre-dose to 72 hours post-dose (each cycle is 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 4 | 7
Hours | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | 10.32 (39.41) | 10.64 (27.39) | NA (NA) — Mean cannot be calculated due to low number participants. | NA (NA) — Mean cannot be calculated due to low number participants. | 6.506 (44.51) | 7.562 (51.64)

7. Secondary Outcome: Accumulation Ratio for Area Under Curve (Rac AUC)
Description: The Rac AUC of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents. Accumulation ratio for AUC, calculated by multiple dose AUCτ/single dose AUC(0-12) or AUC(0-24).
Time Frame: Monotherapy: Cycle 1 Day 8 Pre-dose to 12 hours post dose; Combination therapy: Cycle 1 Days 7 and 8 Pre-dose to 8 hours post dose (each cycle is 28 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Ratio | NA (NA) — Mean cannot be calculated due to low number participant. |  | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. |  |  |  | NA (NA) — Mean cannot be calculated due to low number participants. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant.

8. Secondary Outcome: Accumulation Ratio for Cmax (Rac Cmax)
Description: The Rac Cmax of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents. Accumulation ratio for Cmax, calculated by multiple dose Cmax/single dose Cmax.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 2 | 3 | 2 | 1 | 5
Ratio | NA (NA) — Mean cannot be calculated due to low number participant. |  | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participants. | 1.348 (1.272) | NA (NA) — Mean cannot be calculated due to low number participants. | NA (NA) — Mean cannot be calculated due to low number participants. | 1.157 (23.99)

9. Secondary Outcome: Dose Proportionality (TCP)
Description: The TCP of AZD7648, following a single dose and at steady state after multiple dosing, when given orally as monotherapy and in combination with anti-cancer agents. Temporal change parameter in systemic exposure, calculated as multiple dose AUCtau/single dose AUCinf.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Ratio | NA (NA) — Mean cannot be calculated due to low number participant. |  | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant. |  |  |  | NA (NA) — Mean cannot be calculated due to low number participants. | NA (NA) — Mean cannot be calculated due to low number participant. | NA (NA) — Mean cannot be calculated due to low number participant.

10. Primary Outcome: Number of Patients With Adverse Events or Serious Adverse Events
Description: Safety and tolerability of AZD7648 when given orally to patients with advanced malignancies, as monotherapy and in combination with anti-cancer agents was assessed.
Time Frame: From Screening (Day -28) till study drug discontinuation (3.2 years)
Population: All patients who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 3 | 2 | 2 | 5 | 7
Participants
  Any AE | 0 | 1 | 1 | 1 | 2 | 4 | 3 | 2 | 2 | 4 | 7
  Any AE possibly related to AZD7648 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 4 | 7
  Any AE possibly related to PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE possibly related to PLD |  |  |  |  |  |  |  | 2 | 2 | 4 | 4
  Any AE of CTCAE Grade 3 or higher | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 2 | 2 | 0 | 5
  Any AE of CTCAE Grade 3 or higher, possibly related to AZD7648 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 4
  Any AE of CTCAE Grade 3 or higher, possibly related to PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE of CTCAE Grade 3 or higher, possibly related to PLD |  |  |  |  |  |  |  | 2 | 2 | 0 | 1
  Any AE with outcome of death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Any AE with outcome of death, possibly related to AZD7648 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE with outcome of death, possibly related to PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE with outcome of death, possibly related to PLD |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
  Any SAE | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 0 | 4
  Any SAE, possibly related to AZD7648 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Any SAE, possibly related to PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any SAE, possibly related to PLD |  |  |  |  |  |  |  | 1 | 0 | 0 | 0
  Any SAE with outcome of death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Any SAE with outcome of death, possibly related to AZD7648 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE with outcome of death, possibly related to PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any SAE with outcome of death, possibly related to PLD |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
  Any SAE causing discontinuation of AZD7648 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Any SAE causing discontinuation of AZD7648, possibly related to AZD7648 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any SAE causing discontinuation of AZD7648, possibly related to PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any SAE causing discontinuation of AZD7648, possibly related to PLD |  |  |  |  |  |  |  | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of AZD7648 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1
  Any AE leading to discontinuation of PLD: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE leading to discontinuation of PLD |  |  |  |  |  |  |  | 0 | 1 | 1 | 1
  Any AE leading to AZD7648 dose reduction | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
  Any AE leading to PLD dose reduction: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE leading to PLD dose reduction |  |  |  |  |  |  |  | 0 | 0 | 0 | 1
  Any AE leading to AZD7648 dose interruption | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 4
  Any AE leading to PLD dose interruption: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE leading to PLD dose interruption |  |  |  |  |  |  |  | 2 | 1 | 1 | 4
  Any AE leading to AZD7648 dose modification | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 5
  Any AE leading to PLD dose modification: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 7
  Any AE leading to PLD dose modification |  |  |  |  |  |  |  | 2 | 1 | 1 | 5

11. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as an AE that occurs from the first dose of study treatment up to and including Cycle 1, Day 28 (the DLT assessment period) that is assessed as unrelated to the disease, intercurrent illness, or concomitant medications.
Time Frame: From Screening (Day -28) till study drug discontinuation (3.2 years)
Population: All patients who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 3 | 2 | 2 | 4 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1

12. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients who have a confirmed visit response of complete response (CR) or partial response (PR) prior to any evidence of progression (as defined by Response Evaluation Criteria in Solid Tumours 1.1). CR is defined when all target lesions (TLs) and non-target lesions (NTLs) present at baseline have disappeared (with the exception of lymph nodes which must be <10mm to be considered non pathological) and no new lesions have developed since baseline. PR is defined when the sum of diameters of the TLs has decreased by 30% or more compared to baseline (with no evidence of progression) and the NTLs are at least stable with no evidence of new lesions.
Time Frame: First dose of study treatment on Cycle 1 Day 1 (each cycle is 28 days) until progression or the last evaluable assessment in the absence of progression (3.2 years)
Population: Evaluable for objective response set included all patients who had a measurable baseline disease (having at least one measurable target lesion, not previously irradiated, which is ≥ 10 mm in the longest diameter (LD) (except lymph nodes which must have short axis ≥ 15 mm) by RECIST 1.1 assessment and received at least one dose of any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 4 | 2 | 2 | 2 | 5 | 6
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 0 | 0

13. Secondary Outcome: Progression Free Survival (PFS) for Monotherapy
Description: PFS is defined as the time from first dose of Cycle 1 until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from study therapy or receives another anti-cancer therapy prior to progression. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as increased by > 20% or more compared to the smallest sum of diameters on study.
Time Frame: At 12 months
Population: Evaluable for efficacy set included all patients who received at least 1 dose of any study treatment and have a baseline tumour assessment according to RECIST 1.1.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 3
Months | NA [NA to NA] — Median cannot be calculated due low number of participant. | NA [NA to NA] — Median cannot be calculated due low number of participant. | NA [NA to NA] — Median cannot be calculated due low number of participant. | NA [NA to NA] — Median cannot be calculated due low number of participant. | 1.91 [1.71 to 3.42] | 2.50 [1.64 to 3.52] | 1.51 [1.05 to 7.20]

14. Secondary Outcome: Progression Free Survival (PFS) for Combination Therapy
Description: as for outcome 13
Time Frame: At 18 months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
Number analyzed (Participants) | 2 | 2 | 5 | 7
Months | NA [NA to NA] — Median cannot be calculated due low number of participants. | NA [NA to NA] — Median cannot be calculated due low number of participants. | 1.74 [1.66 to 1.84] | 2.07 [1.87 to 4.11]

ADVERSE EVENTS:
Time Frame: From Screening (Day -28) till study drug discontinuation (3.2 years)
Arm/Group | Cohort 1: AZD7648 Dose A (Monotherapy) | Cohort 2: AZD7648 Dose A1 (Monotherapy) | Cohort 3: AZD7648 Dose B1 (Monotherapy) | Cohort 4: AZD7648 Dose C1 (Monotherapy) | Cohort 5: AZD7648 Dose D1 (Monotherapy) | Cohort 6: AZD7648 Dose E1 (Monotherapy) | Cohort 7: AZD7648 Dose F1 (Monotherapy) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 1/1 | 1/1 | 1/3 | 1/4 | 0/3 | 0/2 | 1/2 | 0/5 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 1/3 | 4/4 | 0/3 | 1/2 | 1/2 | 0/5 | 4/7
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/1 | 1/1 | 2/3 | 4/4 | 3/3 | 2/2 | 2/2 | 4/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1: AZD7648 Dose A (Monotherapy) (N=1) | Cohort 2: AZD7648 Dose A1 (Monotherapy) (N=1) | Cohort 3: AZD7648 Dose B1 (Monotherapy) (N=1) | Cohort 4: AZD7648 Dose C1 (Monotherapy) (N=1) | Cohort 5: AZD7648 Dose D1 (Monotherapy) (N=3) | Cohort 6: AZD7648 Dose E1 (Monotherapy) (N=4) | Cohort 7: AZD7648 Dose F1 (Monotherapy) (N=3) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) (N=2) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) (N=2) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) (N=5) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy) (N=7)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1: AZD7648 Dose A (Monotherapy) (N=1) | Cohort 2: AZD7648 Dose A1 (Monotherapy) (N=1) | Cohort 3: AZD7648 Dose B1 (Monotherapy) (N=1) | Cohort 4: AZD7648 Dose C1 (Monotherapy) (N=1) | Cohort 5: AZD7648 Dose D1 (Monotherapy) (N=3) | Cohort 6: AZD7648 Dose E1 (Monotherapy) (N=4) | Cohort 7: AZD7648 Dose F1 (Monotherapy) (N=3) | Cohort 1: AZD7648 Dose C1 + PLD (Combination Therapy) (N=2) | Cohort 1: AZD7648 Dose C + PLD (Combination Therapy) (N=2) | Cohort 2: AZD7648 Dose C2 + PLD (Combination Therapy) (N=5) | Cohort 3: AZD7648 Dose X + PLD (Combination Therapy) (N=7)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 7 (9)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (9) | 0 (0) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1/3 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 4 (6)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03907969/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT03907969/SAP_001.pdf